CLINICAL TRIAL: NCT01546987
Title: Phase III Trial of Dose Escalated Radiation Therapy and Standard Androgen Deprivation Therapy (ADT) With a GNRH Agonist vs. Dose Escalated Radiation Therapy and Enhanced ADT With a GNRH Agonist and TAK-700 For Men With High Risk Prostate Cancer
Brief Title: Hormone Therapy, Radiation Therapy, and Steroid 17alpha-monooxygenase TAK-700 in Treating Patients With High-Risk Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 1115; CDR0000727326; NCI-2012-00700 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-03-03; First posted 2012-03-07 (Estimated); Results first posted 2023-04-18 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIA prostate cancer; stage IIB prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gonadotropin-Releasing Hormone; Leuprolide; Goserelin; Buserelin; Triptorelin Pamoate; Androgen Antagonists; Flutamide; bicalutamide; orteronel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADT + RT (Active Comparator): Standard androgen deprivation therapy (ADT) beginning two months prior to radiation therapy (RT). ADT comprised of anti-androgen continuing for two years and GnRH agonist stopping at end of RT.
  Interventions: Drug: GnRH agonist; Drug: Anti-androgen; Radiation: Radiation therapy
- TAK-700 + ADT + RT (Experimental): TAK-700 and standard androgen deprivation therapy (ADT) beginning two months prior to radiation therapy (RT). ADT comprised of anti-androgen continuing for two years and GnRH agonist stopping at end of RT. TAK-700 continues for two years.
  Interventions: Drug: GnRH agonist; Drug: Anti-androgen; Drug: TAK-700; Radiation: Radiation therapy

INTERVENTIONS:
Drug: GnRH agonist — LHRH agonists are administered with a variety of techniques. The manufacturer's instructions should be followed. Begins within 6 weeks after registration (if not started prior) at same time as anti-androgen and TAK-700 (if applicable).
  Other Names: LHRH analog; leuprolide; goserelin; buserelin; triptorelin; Gonadotropin-releasing hormone (GnRH) Agonist; LHRH agonist
Drug: Anti-androgen — Starts at same time as GnRH agonist, ends at end of radiation therapy. Either flutamide (orally 250 mg three times a day) or bicalutamide (orally 50 mg once a day).
  Other Names: flutamide; bicalutamide; androgen suppression
Drug: TAK-700 — 300 mg twice daily (BID) (600 mg per day) orally, continuously for 2 years starting with ADT.
  Arms: TAK-700 + ADT + RT
Radiation: Radiation therapy — Starts 8-10 weeks after initiation of ADT. Initially 45 Gy (1.8 Gy / fraction) to prostate and pelvic lymph nodes delivered with 3DCRT/IMRT, then a boost using intensity-modulated radiation therapy (IMRT), low dose rate (LDR) brachytherapy, or high dose rate (HDR) brachytherapy.

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Drugs, such as steroid 17alpha-monooxygenase TAK-700, when used with other hormone therapy, may lessen the amount of androgens made by the body. Radiation therapy uses high energy x rays to kill tumor cells. This may be an effective treatment for prostate cancer when combined with hormone therapy. Studying quality-of-life in patients having cancer treatment may help identify the intermediate- and long-term effects of treatment on patients with prostate cancer.

PURPOSE: This randomized phase III trial is studying the use of hormone therapy, including TAK-700, together with radiation therapy in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the difference in overall survival of patients with clinically localized prostate cancer with unfavorable prognostic features between a) standard treatment (androgen-deprivation therapy [ADT] + radiotherapy) and b) standard treatment with the addition of 24 months of steroid 17alpha-monooxygenase TAK-700 (TAK-700).

Secondary

* To characterize differences between the treatment groups with respect to incidence of unexpected grade ≥ 3 adverse events and/or clinically significant decrement in patient-reported quality of life (QOL) among subjects treated with TAK-700.
* To compare rates and cumulative incidence of biochemical control (freedom from PSA failure), local/regional progression, and distant metastases.
* To compare rate and cumulative incidence of clinical failure, defined as prostate-specific antigen (PSA) > 25 ng/mL, documented local disease progression, regional or distant metastasis, or initiation of ADT.
* To compare prostate cancer-specific survival and other-cause mortality.
* To compare the change in severity of fatigue as measured by the Patient-Reported Outcome Measurement Information System (PROMIS) fatigue short form.
* To compare changes in patient-reported QOL as measured by Expanded Prostate Cancer Index Composite (EPIC).
* To assess quality-adjusted survival using the EQ-5D.
* To compare nadir and average serum testosterone at 12 and 24 months during treatment.
* To compare changes in hemoglobin A1C, fasting glucose, and fasting insulin during 24 months of systemic treatment and during the first three years of follow-up.
* To compare changes in fasting lipid levels during 24 months of treatment and during the first three years of follow-up.
* To compare changes in body mass index (BMI) during 24 months of treatment and during the first three years of follow-up.
* To compare the incidence of adverse events ascertained via CTCAE version 4.
* To compare the rate of recovery of testosterone to > 230 ng/dL (accepted threshold for supplementation) after 12 and 24 months of follow-up.
* To compare the median time to recovery of testosterone to > 230 ng/dL during the first five years of follow-up.
* To assess cumulative incidence of relevant clinical survivorship endpoints including new diagnosis of type 2 diabetes, coronary artery disease, myocardial infarction, stroke, pulmonary embolism, deep vein thrombosis, or osteoporotic fracture.

OUTLINE: This is a multicenter, randomized study. Patients are stratified according to risk group (see Disease Characteristics) and type of radiation therapy (RT) boost (intensity-modulated RT (IMRT) vs brachytherapy). Patients are randomized to 1 of 2 treatment arms.

After completion of study therapy, patients are followed every 3 months for 2 years, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of adenocarcinoma of the prostate within 180 days prior to registration at high risk for recurrence as determined by one of the following combinations:

   * Gleason Score (GS) ≥ 9, PSA ≤ 150 ng/mL, any T stage
   * GS ≥ 8, PSA < 20 ng/mL, T stage ≥ T2
   * GS ≥ 8, PSA ≥ 20-150 ng/mL, any T stage
   * GS ≥ 7, PSA ≥ 20-150 ng/mL, any T stage
2. History/physical examination within 60 days prior to registration.
3. Clinically negative lymph nodes as established by imaging [abdominal and/or pelvic computerized tomography (CT) or abdominal and/or pelvic magnetic resonance imaging (MRI)], nodal sampling, or dissection within 90 days prior to registration.

   •Patients with lymph nodes equivocal or questionable by imaging are eligible if the nodes are < 2.0 cm.
4. No distant metastases (M0) on bone scan within 90 days prior to registration (18F-Na bone scan is an acceptable substitute).

   •Equivocal bone scan findings are allowed if plain films are negative for metastasis.
5. Baseline serum prostate-specific antigen (PSA) value performed with an FDA-approved assay (e.g., Abbott, Hybritech), obtained prior to any luteinizing hormone-releasing hormone (LHRH) or anti-androgen therapy, within 180 days of randomization.
6. Androgen deprivation therapy (ADT), such as LHRH agonists (e.g., goserelin, leuprolide), anti-androgens (e.g., flutamide, bicalutamide), estrogens (e.g., DES), or surgical castration (orchiectomy), may have been started prior to registration, provided that registration is within 50 days of beginning ADT. Please note: If the patient has started ADT he will not be eligible to participate in the quality of life component of this study.
7. Prior testosterone administration is allowed if last administered at least 90 days prior to registration.
8. Zubrod Performance Status 0-1 within 21 days prior to registration
9. Age ≥ 18
10. Complete blood count (CBC)/differential obtained within 14 days prior to registration on study, with adequate bone marrow function defined as follows:

    * Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3
    * Platelets ≥ 100,000 cells/mm3
    * Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.)
11. Serum creatinine < 2.0 mg/dl and creatinine clearance (can be calculated) > 40 mL/minute within 21 days prior to registration
12. Bilirubin < 1.5x upper limit of normal (ULN) and alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5x ULN within 21 days prior to registration
13. Serum testosterone within 21 days prior to registration
14. Chemistry (including sodium, potassium, chloride, bicarbonate (carbon dioxide), blood urea nitrogen (BUN), glucose, calcium, magnesium and phosphorous) and liver panels (including albumin and alkaline phosphatase) obtained within 21 days prior to registration
15. Fasting glucose, fasting insulin, lipid panel [cholesterol, triglyceride, high-density lipoprotein (HDL), low-density lipoprotein (LDL)], and Hemoglobin A1C within 21 days prior to registration
16. Screening calculated ejection fraction of ≥ to institutional lower limit of normal by multiple gated acquisition (MUGA) scan or by echocardiogram (ECHO).
17. Baseline electrocardiogram (ECG) within 180 days prior to registration
18. Patients, even if surgically sterilized (ie, status post vasectomy), who:

    1. Agree to practice effective barrier contraception during the entire study treatment period and for 4 months (120 days) after the last dose of study drug, or
    2. Agree to completely abstain from intercourse.
19. Patient must be able to provide study-specific informed consent prior to study entry.

Exclusion Criteria:

1. PSA > 150
2. Definite evidence of metastatic disease.
3. Pathologically positive lymph nodes or nodes > 2.0 cm on imaging.
4. Prior radical prostatectomy, cryosurgery for prostate cancer, or bilateral orchiectomy for any reason.
5. Prior invasive malignancy (except non-melanoma skin cancer) unless disease-free or not requiring systemic therapy for a minimum of 3 years.
6. Prior systemic chemotherapy for prostate cancer (Note that prior chemotherapy for a different cancer is allowed).
7. Prior radiotherapy, including brachytherapy, to the region of the prostate that would result in overlap of radiation therapy fields.

   •Any patient undergoing brachytherapy must have transrectal ultrasound confirmation of prostate volume <60 cc, American Urological Association (AUA) score ≤15 within 60 days of registration, and no history of prior transurethral resection of the prostate (TURP); prior TURP is permitted for patients who receive external beam radiation therapy [EBRT] only).
8. Previous hormonal therapy for > 50 days.
9. Known hypersensitivity to TAK-700 or related compounds
10. A history of adrenal insufficiency
11. History of myocardial infarction, unstable symptomatic ischemic heart disease, ongoing arrhythmias of Grade > 2 [NCI CTCAE, version 4.02] (U.S. Department of Health and Human Services, National Institutes of Health National Cancer Institute, 2009), thromboembolic events (eg, deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), or any other cardiac condition (e.g., pericardial effusion restrictive cardiomyopathy) within 6 months prior to registration. Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed.
12. New York Heart Association Class III or IV heart failure.
13. ECG abnormalities of:

    1. Q-wave infarction, unless identified 6 or more months prior to screening
    2. QTc interval > 460 msec
14. Patients who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
15. Prior allergic reaction to the drugs involved in this protocol.
16. Study entry PSA obtained during the following time frames:

    1. 10-day period following prostate biopsy;
    2. following initiation of hormonal therapy.
17. Cushing's syndrome
18. Severe chronic renal disease (serum creatinine > 2.0 mg/dl and confirmed by creatinine clearance < 40 mL/minute)
19. Chronic liver disease (bilirubin > 1.5x ULN, ALT or AST > 2.5x ULN)
20. Chronic treatment with glucocorticoids within one year
21. Uncontrolled hypertension despite appropriate medical therapy within 21 days prior to registration (blood pressure of greater than 150 mm Hg systolic and 90 mm Hg diastolic at 2 separate measurements no more than 60 minutes apart during Screening visit)
22. Unwilling or unable to comply with the protocol or cooperate fully with the investigator and site personnel.
23. Major surgery within 14 days prior to registration
24. Serious infection within 14 days prior to registration
25. Uncontrolled nausea, vomiting, or diarrhea [Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3] despite appropriate medical therapy at the time of registration
26. Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of TAK-700, including difficulty swallowing tablets

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2025-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Dror Michaelson, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (172):
- United States (165):
  - The Kirklin Clinic at Acton Road, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Oncology-Deer Valley Center, Phoenix, Arizona
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Veterans Administration Long Beach Medical Center, Long Beach, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - University of Southern California/Norris Cancer Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - University of California At San Diego, San Diego, California
  - UCSF-Mount Zion, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Stanford University Hospitals and Clinics, Stanford, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center, Vallejo, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Poudre Valley Radiation Oncology, Fort Collins, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - William Backus Hospital, Norwich, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - University of Miami Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Grady Health System, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Saint Joseph's-Candler Health System, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Idaho Urologic Institute PA, Meridian, Idaho
  - Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Hines Veterans Administration Hospital, Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kansas City Cancer Centers-Southwest, Overland Park, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Touro Infirmary, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Saint Agnes Hospital, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Saint Anne's Hospital, Fall River, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - North Shore Medical Center Cancer Center, Peabody, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - McLaren-Flint, Flint, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Great Lakes Cancer Institute-Lapeer Campus, Lapeer, Michigan
  - McLaren Cancer Institute-Owosso, Owosso, Michigan
  - Northern Michigan Regional Hospital, Petoskey, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center - Saint Peters, City of Saint Peters, Missouri
  - Kansas City Cancer Center - South, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Kansas City Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - The Nebraska Medical Center, Omaha, Nebraska
  - Concord Hospital, Concord, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Geaugra Hospital, Chardon, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Summa Health Center at Lake Medina, Medina, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center Ireland Cancer Center, Middleburg Heights, Ohio
  - UHHS-Chagrin Highlands Medical Center, Orange, Ohio
  - Robinson Radiation Oncology, Ravenna, Ohio
  - Ireland Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Flower Hospital, Sylvania, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Rogue Valley Medical Center, Medford, Oregon
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - The Regional Cancer Center, Erie, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Texas Oncology PA - Bedford, Bedford, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The Klabzuba Cancer Center, Fort Worth, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Texas Cancer Center-Sherman, Sherman, Texas
  - Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Intermountain Medical Center, Murray, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Sentara Hospitals, Norfolk, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Roanoke, Virginia
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - Saint Francis Hospital, Federal Way, Washington
  - Virginia Mason CCOP, Seattle, Washington
  - Appleton Medical Center, Appleton, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran, La Crosse, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia Saint Mary's Water Tower Medical Commons, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Clement J. Zablocki VA Medical Center, Milwaukee, Wisconsin
  - Wheaton Franciscan Cancer Care - All Saints, Racine, Wisconsin
  - Door County Cancer Center, Sturgeon Bay, Wisconsin
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA-Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - London Regional Cancer Program, London, Ontario
  - Ottawa Health Research Institute-General Division, Ottawa, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Started | 118 | 120
Eligible | 115 | 116
Eligible Participants Who Consented to Quality of Life (QOL) Component | 103 | 94
Completed | 115 | 116
Not Completed | 3 | 4
Not completed — Protocol Violation | 3 | 4

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | ADT + RT | TAK-700 + ADT + RT | Total
Number analyzed (Participants) | 115 | 116 | 231
Age, Customized [Count of Participants; unit: Participants]
  ≤ 49 years | 2 | 1 | 3
  50 - 59 years | 16 | 22 | 38
  60 - 69 years | 44 | 41 | 85
  ≥ 70 years | 53 | 52 | 105
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 115 | 116 | 231
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 111 | 109 | 220
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 10 | 24
  White | 93 | 101 | 194
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 4 | 10
Zubrod Performance Status [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound; 5 = Death.
  Participants
    0 | 99 | 104 | 203
    1 | 16 | 12 | 28
Gleason Score [Count of Participants; unit: Participants] — Gleason score describes prostate cancer based on how abnormal the cancer cells in a biopsy sample look under a microscope. Cells are scored 1-5 with 1 indicating "low-grade" looking similar to normal cells and 5 indicating "high-grade" barely resembling normal cells due to mutation. A pathologist assigns a Gleason grade to the first and second most predominant patterns in the biopsy. The two grades are added together to calculate the Gleason score (between 2 and 10). Cancers with lower scores tend to be less aggressive, while cancers with higher scores end to be more aggressive.
  Participants
    7 | 16 | 18 | 34
    8 | 37 | 30 | 67
    ≥9 | 62 | 68 | 130
Study Entry PSA [Count of Participants; unit: Participants] — Prostate-specific antigen (PSA) is a protein made by the prostate gland and found in the blood. PSA blood levels may be higher than normal in men who have prostate cancer, benign prostatic hyperplasia (BPH), or infection or inflammation of the prostate gland, and are often used to monitor patients who have been treated for prostate cancer to see if their cancer has recurred.
  Participants
    < 20.0 ng/ml | 75 | 75 | 150
    20.0-150.0 ng/ml | 40 | 41 | 81
T-Stage [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 7th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b.
  Participants
    T1a-T1c | 22 | 23 | 45
    T2-T2c | 66 | 58 | 124
    T3-T3b | 24 | 33 | 57
    T4 | 3 | 2 | 5
Risk Factors [Count of Participants; unit: Participants]
  Gleason ≥ 9, PSA ≤150, any T-stage | 65 | 67 | 132
  Gleason 8, PSA <20, and ≥T2 | 23 | 21 | 44
  Gleason 8, PSA ≥20-150, any T-stage | 13 | 10 | 23
  Gleason 7, PSA ≥20-150, any T-stage | 14 | 18 | 32
N-Stage N0 [Count of Participants; unit: Participants] — Regional lymph nodes staging per American Joint Committee on Cancer (AJCC) 7th ed. refers to the number and/or extent of spread of lymph nodes that contain cancer. N0 means lymph nodes aren't involved. A higher number means the cancer is in more lymph nodes, farther away from the original tumor. NX means the lymph nodes cannot be assessed.
  Participants | 115 | 116 | 231
M-Stage M0 [Count of Participants; unit: Participants] — Metastasis stage per the American Joint Committee on Cancer (AJCC) 7th ed. refers to the spread of the cancer to organs and tissues in other parts of the body. M0 = No distant metastasis; M1 = Distant metastasis; MX = Distant metastasis cannot be assessed.
  Participants | 115 | 116 | 231
ADT Started Prior to Registration [Count of Participants; unit: Participants] — Population: Trial was amended midstudy to add this stratification variable, therefore data was not collected on all participants.
  Participants
    number analyzed (Participants) | 42 | 45 | 87
    No | 31 | 25 | 56
    Yes | 11 | 20 | 31
RT Boost Modality [Count of Participants; unit: Participants]
  Intensity-modulated radiation therapy (IMRT) | 103 | 105 | 208
  Low dose rate (LDR) permanent prostate implant (PPI) | 12 | 10 | 22
  High dose rate (HDR) implant | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Biochemical Failure (Primary Endpoint of Revised Protocol)
Description: Note, the revised protocol (see Limitations and Caveats) changed this outcome measure from secondary (original protocol) to primary. Biochemical failure will be defined by the Phoenix definition (PSA ≥ 2 ng/ml over the nadir PSA, the presence of local, regional, or distant recurrence, or the initiation of salvage androgen deprivation therapy. Time to failure is defined as time from randomization to the date of first failure, last known follow-up (censored), or death without failure (competing risk). Failure rates are estimated using the cumulative incidence method, while treatment effect comparisons are based on cause-specific hazards (deaths censored). Five-year rates are provided here.
Time Frame: From randomization to last follow-up. Follow-up schedule: every 3 months from start of treatment for 2 years, then every 6 months for 3 years, then yearly. Maximum follow-up at time of analysis was 9.1 years. Five-year rates are reported here.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 115 | 116
percentage of participants | 17.3 [10.7 to 25.2] | 12.8 [7.1 to 20.1]
Statistical Analysis 1: Comparison: ADT + RT vs TAK-700 + ADT + RT; Revised protocol due to early accrual closure (September 2014) computes that seventy events with five years of additional follow-up after early accrual closure provides 70% power (at one-sided alpha = 0.05) to detect a 40% reduction in the assumed rate control arm rate of is 0.08/year; Test type: Superiority; p = 0.55, Log Rank — One-sided significance level = 0.05; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.47 to 1.48] — Reference level = ADT + RT

2. Secondary Outcome: Percentage of Patients Alive [Overall Survival] (Primary Endpoint of Original Protocol)
Description: Note, the revised protocol (see Limitations and Caveats) changed this outcome measure from primary (original protocol) to secondary. Overall survival time is defined as time from randomization to the date of death from any cause or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. 5-year rates are provided.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 115 | 116
percentage of participants | 89.4 [83.5 to 95.3] | 88.1 [81.8 to 94.4]
Statistical Analysis 1: Comparison: ADT + RT vs TAK-700 + ADT + RT; Revised protocol due to early accrual closure (September 2014) computes that 5-year survival of 78% and annual hazard rate of 0.055 for ADT + RT arm, with five years of additional follow-up after early accrual closure provides 28% power (at two-sided alpha = 0.05) to detect a 33% reduction in failure rate; Test type: Superiority; p = 0.27, Log Rank — Two-sided significance level = 0.05; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.38 to 1.31] — Reference level = ADT + RT

3. Secondary Outcome: Percentage of Participants With Grade 3 or Higher Adverse Events
Description: Time to grade 3 or higher adverse event (event) is defined as time from randomization to the date of first event, last known follow-up (censored), or death without failure (competing risk). Event rates are estimated using the cumulative incidence method, while treatment effect comparisons are based on cause-specific hazards (deaths censored). Five-year rates are provided here.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 115 | 116
percentage of participants | 34.9 [26.0 to 43.9] | 58.9 [48.8 to 67.6]
Statistical Analysis 1: Comparison: ADT + RT vs TAK-700 + ADT + RT; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 2.29, 95% CI 2-sided [1.54 to 3.40] — Reference level = ADT + RT arm

4. Secondary Outcome: Percentage of Participants With Local Progression
Description: Local recurrence (failure) is defined as biopsy proven recurrence within the prostate gland. Time to failure is defined as time from randomization to the date of failure, last known follow-up (censored), or death without failure (competing risk). Failure rates are estimated using the cumulative incidence method, while treatment effect comparisons are based on cause-specific hazards (deaths censored). Five-year rates are provided here.
Time Frame: From randomization to last follow-up. Follow-up schedule: every 3 months from start of treatment for 2 years, then every 6 months for 3 years, then yearly. Maximum follow-up at time of analysis was 9.1 years. Five-year rates reported.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 115 | 116
percentage of participants | 2.9 [0.8 to 7.6] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: ADT + RT vs TAK-700 + ADT + RT; Test type: Superiority; p = 0.99, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.33 to 3.13]

5. Secondary Outcome: Percentage of Participants With Distant Metastases
Description: Distant metastases (failure) is defined as imaging or biopsy demonstrated evidence for systemic recurrence. Biopsy was not required, however it was encouraged in absence of a rising PSA. Time to failure is defined as time from randomization to the date of first failure, last known follow-up (censored), or death without failure (competing risk). Failure rates are estimated using the cumulative incidence method, while treatment effect comparisons are based on cause-specific hazards (deaths censored). Five-year rates are provided here. Note, the protocol lists this endpoint as regional or distant metastasis, but regional progression data was not collected.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 115 | 116
percentage of participants | 6.8 [3.0 to 12.7] | 2.9 [0.8 to 7.7]
Statistical Analysis 1: Comparison: ADT + RT vs TAK-700 + ADT + RT; Revised protocol due to early accrual closure (September 2014) computes that 5-year survival of 78% and annual hazard rate of 0.02 for ADT + RT arm, with five years of additional follow-up after early accrual closure provides 32% power (at two-sided alpha = 0.05) to detect a 50% reduction in failure rate; Test type: Superiority; p = 0.48, Log Rank — Two-sided significance level = 0.05; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.29 to 1.75] — Reference level = ADT + RT arm

6. Secondary Outcome: Percentage of Participants With General Clinical Treatment Failure
Description: General clinical treatment failure (GCTF) is defined as: PSA > 25 ng/ml, documented local disease progression, regional or distant metastasis, or initiation of salvage androgen deprivation therapy. Failure time is defined as time from registration to the date of failure, last known follow-up (censored), or death without failure (competing risk). Failure rates are estimated using the cumulative incidence method, while treatment effect comparisons are based on cause-specific hazards (deaths censored). Five-year rates are provided here.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 115 | 116
percentage of participants | 12.5 [7.0 to 19.6] | 6.8 [3.0 to 12.8]
Statistical Analysis 1: Comparison: ADT + RT vs TAK-700 + ADT + RT; Test type: Superiority; p = 0.65, Log Rank — Two-sided significance level = 0.05; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.45 to 1.63] — Reference level = ADT + RT

7. Secondary Outcome: Percentage of Participants With Death Due to Prostate Cancer
Description: Time to prostate cancer death is defined as time from randomization to the date of death due to prostate cancer, last known follow-up (censored), or death due to other causes (competing risk). Failure rates were to be estimated using the cumulative incidence method. If too few events occur for meaningful estimates, then only counts of events will be reported.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 115 | 116
percentage of participants | 7.7 [3.6 to 13.9] | 4.9 [1.8 to 10.5]

8. Secondary Outcome: Change in Patient-Reported Outcome Measurement Information System (PROMIS) Fatigue Short Form at One Year
Description: The PROMIS Fatigue short form 8a contains 8 questions, each with 5 responses ranging from 1 to 5, evaluating self-reported fatigue symptoms over the past 7 days. The total score is the sum of all questions which is then converted into a pro-rated T-score with a mean of 50 and standard deviation of 10, with a possible range of 33.1 to 77.8. Higher scores indicate more fatigue. Change is defined as value at one year - value at baseline. Positive change from baseline indicates increased fatigue at one year.
Time Frame: Baseline, one year
Population: Eligible participants who consented to quality of life component and had baseline and one-year data.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 78 | 73
T-score | 2.78 (7.21) | 3.16 (8.24)
Statistical Analysis 1: Comparison: ADT + RT vs TAK-700 + ADT + RT; One hundred thirty evaluable participants (arms combined), provides 81% power to detect a moderate effect size of 0.5 using a two-sample test of the difference in means with a two-sided type I error of 0.05; Test type: Superiority; p = 0.76, t-test, 2 sided

9. Secondary Outcome: Change in Patient-reported Quality of Life as Measured by Expanded Prostate Cancer Index Composite (EPIC) Short Form at One Year
Description: The EPIC-Short Form is a 26-item, validated self-administered tool to assess disease-specific aspects of prostate cancer and its therapies consisting of five summary domains (bowel, urinary incontinence, urinary irritation/obstruction, sexual, and hormonal function). Responses for each item form a Likert scale which are transformed to a 0-100 scale. A domain score is the average of the transformed domain item scores, ranging from 0-100 with higher scores representing better health-related quality of life (HRQOL). Change at one year is defined as one-year value - baseline value. Positive change at one year indicates improved quality of life.
Time Frame: Baseline, one year
Population: Eligible participants with data for any of the four domains.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 102 | 94
score on a scale
  Bowel domain: number analyzed (Participants) | 78 | 70
  Bowel domain | -5.45 (9.10) | -7.04 (15.50)
  Urinary domain: number analyzed (Participants) | 77 | 71
  Urinary domain | -1.67 (13.90) | -5.31 (15.46)
  Sexual domain: number analyzed (Participants) | 72 | 67
  Sexual domain | -24.18 (27.64) | -27.26 (25.98)
  Hormonal domain: number analyzed (Participants) | 77 | 72
  Hormonal domain | -17.31 (15.36) | -17.45 (16.59)
Statistical Analysis 1: Comparison: ADT + RT vs TAK-700 + ADT + RT; [Bowel domain] One hundred thirty evaluable participants (arms combined), provides 81% power to detect a moderate effect size of 0.5 using a two-sample test of the difference in means with a two-sided type I error of 0.05; Test type: Superiority; p = 0.44, t-test, 2 sided
Statistical Analysis 2: Comparison: ADT + RT vs TAK-700 + ADT + RT; [Urinary domain] One hundred thirty evaluable participants (arms combined), provides 81% power to detect a moderate effect size of 0.5 using a two-sample test of the difference in means with a two-sided type I error of 0.05; Test type: Superiority; p = 0.13, t-test, 2 sided
Statistical Analysis 3: Comparison: ADT + RT vs TAK-700 + ADT + RT; [Sexual domain] One hundred thirty evaluable participants (arms combined), provides 81% power to detect a moderate effect size of 0.5 using a two-sample test of the difference in means with a two-sided type I error of 0.05; Test type: Superiority; p = 0.50, t-test, 2 sided
Statistical Analysis 4: Comparison: ADT + RT vs TAK-700 + ADT + RT; [Hormonal domain] One hundred thirty evaluable participants (arms combined), provides 81% power to detect a moderate effect size of 0.5 using a two-sample test of the difference in means with a two-sided type I error of 0.05; Test type: Superiority; p = 0.96, t-test, 2 sided

10. Secondary Outcome: Serum Testosterone
Time Frame: Baseline,12 months, 24 months
Population: Eligible participants with data at any of the timepoints.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 115 | 116
ng/dL
  Baseline: number analyzed (Participants) | 98 | 106
  Baseline | 355.75 (225.65) | 357.73 (217.26)
  12 months: number analyzed (Participants) | 67 | 58
  12 months | 35.68 (68.39) | 25.22 (67.49)
  24 months: number analyzed (Participants) | 59 | 116
  24 months | 86.47 (182.40) | 17.36 (32.71)

11. Secondary Outcome: Fasting Total Cholesterol
Time Frame: Baseline, 12 months, 24 months
Population: Eligible participants with data at any of the timepoints.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 114 | 116
mg/dL
  Baseline: number analyzed (Participants) | 100 | 107
  Baseline | 149.71 (68.20) | 154.20 (71.05)
  12 months: number analyzed (Participants) | 82 | 81
  12 months | 160.27 (73.22) | 154.74 (70.85)
  24 months: number analyzed (Participants) | 70 | 67
  24 months | 163.20 (168.63) | 160.61 (77.55)

12. Secondary Outcome: Serum High-density Lipoprotein (HDL)
Time Frame: Baseline, 12 months, 24 months
Population: Eligible participants with data at any of the timepoints.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 114 | 116
mg/dL
  Baseline: number analyzed (Participants) | 101 | 106
  Baseline | 40.91 (20.96) | 41.32 (20.93)
  12 months: number analyzed (Participants) | 80 | 81
  12 months | 44.94 (24.21) | 44.50 (24.21)
  24 months: number analyzed (Participants) | 70 | 67
  24 months | 42.16 (23.77) | 44.85 (23.36)

13. Secondary Outcome: Serum High-density Lipoprotein (LDL)
Time Frame: Baseline, 12 months, 24 months
Population: Eligible participants with data at any of the timepoints.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 114 | 116
mg/dL
  Baseline: number analyzed (Participants) | 100 | 105
  Baseline | 88.78 (45.64) | 87.85 (47.33)
  12 months: number analyzed (Participants) | 77 | 78
  12 months | 86.18 (47.11) | 83.73 (46.86)
  24 months: number analyzed (Participants) | 69 | 64
  24 months | 81.35 (47.73) | 95.34 (59.22)

14. Secondary Outcome: Hemoglobin A1c
Time Frame: Baseline, 12 months, 24 months
Population: Eligible participants with data at any of the timepoints.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 114 | 115
g/dL
  Baseline: number analyzed (Participants) | 103 | 107
  Baseline | 6.12 (1.05) | 6.01 (1.05)
  12 months: number analyzed (Participants) | 73 | 74
  12 months | 6.33 (1.18) | 5.95 (0.73)
  24 months: number analyzed (Participants) | 75 | 70
  24 months | 6.30 (1.59) | 6.04 (0.76)

15. Secondary Outcome: Fasting Plasma Glucose
Time Frame: Baseline, 12 months, 24 months
Population: Eligible participants with data at any of the timepoints.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 112 | 115
mg/dL
  Baseline: number analyzed (Participants) | 112 | 114
  Baseline | 98.99 (51.87) | 100.52 (45.54)
  12 months: number analyzed (Participants) | 91 | 87
  12 months | 102.27 (53.06) | 117.39 (118.40)
  24 months: number analyzed (Participants) | 77 | 76
  24 months | 104.24 (67.43) | 105.51 (40.53)

16. Secondary Outcome: Fasting Plasma Insulin
Time Frame: Baseline, 12 months, 24 months
Population: This data was not collected.
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Body Mass Index (BMI) is a person's weight in kilograms (or pounds) divided by the square of height in meters (or feet). Change from baseline = time point value - baseline value.
Time Frame: Baseline and yearly to five years.
Population: Eligible participants data at baseline and data at any of the post-baseline timepoints.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 111 | 107
kg/m^2
  1 year: number analyzed (Participants) | 97 | 95
  1 year | 0.64 (2.19) | -0.84 (4.28)
  2 years: number analyzed (Participants) | 96 | 88
  2 years | 0.67 (3.76) | -0.34 (2.55)
  3 years: number analyzed (Participants) | 85 | 81
  3 years | 0.75 (3.90) | 0.25 (2.32)
  4 years: number analyzed (Participants) | 78 | 76
  4 years | -0.02 (6.95) | 0.46 (2.70)
  5 years: number analyzed (Participants) | 70 | 71
  5 years | -0.52 (3.01) | 0.15 (2.71)

18. Secondary Outcome: Number of Participants by Highest Grade Adverse Event
Description: Common Terminology Criteria for Adverse Events (version 4.0) grades adverse event severity from 1=mild to 5=death. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data
Time Frame: From registration to last follow-up. Follow-up schedule: every 3 months from start of treatment for 2 years, then every 6 months for 3 years, then yearly. Maximum follow-up at time of analysis was 9.1 years. Five-year rates are reported here.
Population: Eligible participants who started protocol treatment
Measure: Count of Participants; unit: Participants
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 112 | 115
Participants
  Grade 1 | 17 | 2
  Grade 2 | 54 | 45
  Grade 3 | 31 | 55
  Garde 4 | 4 | 9
  Grade 5 | 3 | 1

19. Secondary Outcome: Testosterone Recovery at 12 and 24 Months
Description: Testosterone recovery is defined as testosterone level after treatment greater than 230 ng/dL. Time to testosterone recovery is defined as time from randomization to the date of testosterone recovery, biochemical, local, or distant failure (competing risk), salvage therapy (competing risk), death (competing risk), or last known follow-up (censored). Testosterone recovery rates are estimated using the cumulative incidence method.
Time Frame: From registration to last follow-up. Follow-up schedule: every 3 months from start of treatment for 2 years, then every 6 months for 3 years, then yearly. Maximum follow-up at time of analysis was 9.1 years.
Population: Eligible participants with testosterone data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 112 | 113
percentage of participants
  12 months | 19.4 [12.5 to 27.3] | 12.5 [7.0 to 19.6]
  24 months | 32.9 [24.1 to 41.9] | 17.4 [10.8 to 25.4]

20. Secondary Outcome: Median Testosterone Recovery Time
Description: Testosterone recovery is defined as testosterone level after treatment greater than 230 ng/dL. Testosterone recovery rates are estimated using the Kaplan-Meier method, censoring for biochemical, local, or distant failure, salvage therapy, death, and otherwise alive without event. Testosterone recovery time is defined as time from randomization to testosterone recovery or censoring.
Time Frame: as for outcome 1
Population: Eligible participants with testosterone data
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 112 | 113
years | NA [4.2 to NA] — The median and the upper confidence limit were not reached. | NA [NA to NA] — The median, and the lower and upper 95% confidence limits were not reached
Statistical Analysis 1: Comparison: ADT + RT vs TAK-700 + ADT + RT; Test type: Superiority; p = 0.0104, Log Rank; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.29 to 0.89] — Reference arm = ADT + RT arm

21. Secondary Outcome: Number of Patients With Clinical Survivorship Events
Description: Clinical survivorship events are defined as the following newly diagnosed non-fatal cardiovascular events or other clinical endpoints relevant to prostate cancer survivorship:
  type 2 diabetes, coronary artery disease, myocardial infarction, stroke, pulmonary embolism, deep vein thrombosis, and osteoporotic fracture.
Time Frame: as for outcome 1
Population: Eligible participants
Measure: Count of Participants; unit: Participants
Arm/Group | ADT + RT | TAK-700 + ADT + RT
Number analyzed (Participants) | 115 | 116
Participants
  Type 2 diabetes | 30 | 18
  Coronary artery disease | 16 | 14
  Myocardial infarction | 6 | 8
  Stroke | 5 | 6
  Pulmonary embolism | 10 | 5
  Deep vein thrombosis | 8 | 7
  Osteoporotic fracture | 6 | 1

ADVERSE EVENTS:
Time Frame: From randomization to last follow-up. Follow-up schedule: every 3 months from start of treatment for 2 years, then every 6 months for 3 years, then yearly. Maximum follow-up at time of analysis was 9.1 years.
Description: All-cause mortality was assessed in eligible participants. Adverse events were assessed in eligible participants who started protocol treatment.
Arm/Group | ADT + RT | TAK-700 + ADT + RT
All-Cause Mortality (participants affected / at risk) | 24/115 | 19/116
Serious Adverse Events (participants affected / at risk) | 19/112 | 38/115
Other Adverse Events (participants affected / at risk) | 108/112 | 112/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADT + RT (N=112) | TAK-700 + ADT + RT (N=115)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 1
Aortic valve disease (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 3
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac disorders - Other (Cardiac disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Heart failure (Cardiac disorders) | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 3 | 4
Sinus bradycardia (Cardiac disorders) | 0 | 1
Eye disorders - Other (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Rectal fistula (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Death NOS (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 2
Irritability (General disorders) | 0 | 1
Sudden death NOS (General disorders) | 1 | 0
Gallbladder pain (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Amnesia (Nervous system disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2
Nervous system disorders - Other (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 1 | 3
Syncope (Nervous system disorders) | 2 | 0
Transient ischemic attacks (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Bladder spasm (Renal and urinary disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 2 | 1
Renal calculi (Renal and urinary disorders) | 0 | 3
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1
Hot flashes (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 3
Vascular disorders - Other (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ADT + RT (N=112) | TAK-700 + ADT + RT (N=115)
Anemia (Blood and lymphatic system disorders) | 20 | 23
Abdominal pain (Gastrointestinal disorders) | 8 | 17
Constipation (Gastrointestinal disorders) | 23 | 32
Diarrhea (Gastrointestinal disorders) | 61 | 69
Dyspepsia (Gastrointestinal disorders) | 2 | 6
Fecal incontinence (Gastrointestinal disorders) | 4 | 6
Flatulence (Gastrointestinal disorders) | 11 | 11
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 7
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 18 | 23
Hemorrhoids (Gastrointestinal disorders) | 7 | 6
Nausea (Gastrointestinal disorders) | 9 | 38
Proctitis (Gastrointestinal disorders) | 18 | 13
Rectal hemorrhage (Gastrointestinal disorders) | 17 | 13
Vomiting (Gastrointestinal disorders) | 4 | 16
Edema limbs (General disorders) | 9 | 17
Fatigue (General disorders) | 72 | 91
General disorders and administration site conditio (General disorders) | 9 | 15
Pain (General disorders) | 15 | 18
Infections and infestations - Other (Infections and infestations) | 7 | 4
Urinary tract infection (Infections and infestations) | 7 | 11
Dermatitis radiation (Injury, poisoning and procedural complications) | 4 | 6
Alanine aminotransferase increased (Investigations) | 10 | 25
Alkaline phosphatase increased (Investigations) | 9 | 10
Aspartate aminotransferase increased (Investigations) | 10 | 24
Cholesterol high (Investigations) | 3 | 16
Creatinine increased (Investigations) | 10 | 16
Investigations - Other (Investigations) | 8 | 14
Lymphocyte count decreased (Investigations) | 11 | 10
Weight gain (Investigations) | 10 | 7
Weight loss (Investigations) | 10 | 28
White blood cell decreased (Investigations) | 5 | 13
Anorexia (Metabolism and nutrition disorders) | 10 | 27
Dehydration (Metabolism and nutrition disorders) | 1 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 33 | 39
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 7
Hypertriglyceridemia (Metabolism and nutrition disorders) | 10 | 13
Hypokalemia (Metabolism and nutrition disorders) | 5 | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 10
Hyponatremia (Metabolism and nutrition disorders) | 6 | 11
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 9 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 15
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 15
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 13 | 19
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 6 | 4
Musculoskeletal and connective tissue disorder - (Musculoskeletal and connective tissue disorders) | 11 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 14
Dizziness (Nervous system disorders) | 12 | 29
Dysgeusia (Nervous system disorders) | 2 | 9
Headache (Nervous system disorders) | 10 | 21
Memory impairment (Nervous system disorders) | 6 | 2
Nervous system disorders - Other (Nervous system disorders) | 3 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 8
Anxiety (Psychiatric disorders) | 7 | 14
Depression (Psychiatric disorders) | 13 | 20
Insomnia (Psychiatric disorders) | 19 | 22
Libido decreased (Psychiatric disorders) | 15 | 14
Cystitis noninfective (Renal and urinary disorders) | 14 | 17
Hematuria (Renal and urinary disorders) | 17 | 15
Renal and urinary disorders - Other (Renal and urinary disorders) | 42 | 46
Urinary frequency (Renal and urinary disorders) | 74 | 83
Urinary incontinence (Renal and urinary disorders) | 27 | 18
Urinary retention (Renal and urinary disorders) | 22 | 24
Urinary tract obstruction (Renal and urinary disorders) | 7 | 8
Urinary tract pain (Renal and urinary disorders) | 20 | 21
Urinary urgency (Renal and urinary disorders) | 49 | 37
Erectile dysfunction (Reproductive system and breast disorders) | 49 | 47
Gynecomastia (Reproductive system and breast disorders) | 8 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 | 25
Respiratory, thoracic and mediastinal disorders - (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 9
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 5 | 13
Hot flashes (Vascular disorders) | 83 | 89
Hypertension (Vascular disorders) | 18 | 37
Hypotension (Vascular disorders) | 2 | 6
Vascular disorders - Other (Vascular disorders) | 6 | 6

LIMITATIONS AND CAVEATS:
This study closed to accrual early at 238 participants out of 900 planned due to discontinuation of support from the industry partner (Takeda/Millenium) for further development of TAK-700 in prostate cancer. The study endpoints and statistical considerations were revised to take the smaller sample size into account. The revised protocol contains both the original and revised statistical sections.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT01546987/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT01546987/ICF_001.pdf